CLINICAL TRIAL: NCT00816907
Title: Metformin in the Treatment of Antipsychotic-Induced Weight Gain in Schizophrenia (METS) - Pilot Study
Brief Title: The Use of Metformin in the Treatment of Antipsychotic-Induced Weight Gain in Schizophrenia (The METS Study)
Acronym: METS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01 MH090001-03; N01MH90001 DSIR AT (Other: National Institute of Mental Health); N01MH90001 (NIH); N01MH090001 (NIH)
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Encapsulated metformin 1000-2000 mg/day
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Matching placebo capsules 2-4 daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 500 mg to 1,000 mg taken twice daily for 16 weeks
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — 1 to 2 placebo capsules taken twice daily for 16 weeks
  Arms: Placebo

SUMMARY:
This study will test the usefulness of the medication metformin in treating people with schizophrenia or schizoaffective disorder who are overweight and also taking antipsychotic medications.

DETAILED DESCRIPTION:
Schizophrenia is a chronic mental disorder that is characterized, in part, by psychotic symptoms. Psychotic symptoms include hallucinations and delusions, in which a person has abnormal experiences or beliefs, and are commonly treated with antipsychotic medications. Unfortunately, a side effect of many antipsychotics is unwanted weight gain, which can lead to physical illness. Use of the drug metformin has resulted in weight loss among diabetics. Metformin has also been shown to cause weight loss in preliminary studies of people taking atypical antipsychotics-a newer, second generation of antipsychotic medications. Metformin is currently approved by the Food and Drug Administration to treat only people with diabetes. This study will test the usefulness of prescribing metformin as a second medication to treat people with schizophrenia or schizoaffective disorder who are overweight and taking antipsychotics. The study will also provide important feasibility information for future larger studies.

Participation in this study will last 16 weeks. After undergoing baseline assessments, participants will be randomly assigned to receive either metformin or placebo, both of which will be taken twice daily for the duration of the study. All participants will also receive behavioral therapy that will teach them about reducing their weight through diet and exercise. Participants will undergo assessments at 11 study visits: the first 2 will include screening and baseline testing, the next 2 visits will take place after the first and second weeks of receiving treatment, and the last 7 visits will take place every 2 weeks until the end of the study. Assessments will include measurements of body weight, waist-to-hip ratio, and vital signs; clinical interviews about medication adherence, side effects, and alcohol use; and monthly blood tests to assess levels of lipids, glucose, insulin, and hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of schizophrenia or schizoaffective disorder, as defined by DSM-IV-TR criteria and confirmed by the Structured Clinical Interview for DSM-IV (SCID)
* Duration of illness greater than 1 year, as defined by having initiated antipsychotic treatment at least 1 year prior to study entry
* Adequate decisional capacity to make a choice about participating in this research study
* Body mass index (BMI) at or greater than 27
* Currently being treated with one or a combination of two antipsychotic medications (typical or atypical) and on that drug regimen for at least 2 months prior to study entry, with stable dosages for at least 1 month
* If taking antidepressants, mood stabilizers, or anxiolytics, the dose must be stable for at least 1 month prior to study entry
* Willing to use an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study. Acceptable methods include oral, injectable, or implanted contraceptives; intrauterine devices or barrier methods such as condoms; and diaphragms and spermicides.

Exclusion Criteria:

* Inpatient status
* Clinical Global Impression Severity (CGI-S) score greater than 6
* Currently being treated with more than two antipsychotic medications
* Fasting glucose greater than 125
* Diagnosis of diabetes mellitus or treatment with insulin or oral hypoglycemics
* Previous or current treatment with metformin
* Diagnosis of congestive heart failure
* Renal impairment, as defined by a serum creatinine level greater than 1.5 in males or greater than 1.4 in females, or creatinine estimated glomerular filtration rate (GFR) outside of normal limits
* Hepatic disease, as defined by aspartate transaminase (AST), alanine transaminase (ALT), or c-glutamyl transferase (CGT) greater than 1.5 times upper limit of normal (ULN), or total bilirubin greater than 1.2 times ULN
* Metabolic acidosis, as defined by serum carbon dioxide less than the lower limit of normal
* Known hypersensitivity to metformin
* Pregnant or breastfeeding
* Recent (in the past 30 days) or scheduled radiological studies involving iodinated contrast material
* Alcohol abuse or dependence within the past month, as determined by the SCID
* Other serious and unstable medical condition in the judgment of the investigator
* Diagnosis of mental retardation, delirium, or dementia, as defined by DSM-IV-TR
* Failed to discontinue 4 weeks prior to study entry any medication used for weight loss
* Concurrent treatment with certain drugs that are known to increase metformin blood levels should be discussed with the Project Medical Officer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Fredrik Jarskog, MD, Principal Investigator — Columbia University; Jeffrey A. Lieberman, MD, Principal Investigator — Columbia University; T. Scott Stroup, MD, MPH, Principal Investigator — Columbia University
Locations (16):
- United States (16):
  - Stanford University, Palo Alto, California
  - Mental Health Advocates, Boca Raton, Florida
  - University of Iowa, Iowa City, Iowa
  - Clinical Research Institute, Wichita, Kansas
  - Clinical Insights, Glen Burnie, Maryland
  - Freedom Trail Clinic, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Minnesota School of Medicine, Minneapolis, Minnesota
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - Research Foundation for Mental Hygiene, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University Schizophrenia Research, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Wang B, Ogburn EL, Rosenblum M. Analysis of covariance in randomized trials: More precision and valid confidence intervals, without model assumptions. Biometrics. 2019 Dec;75(4):1391-1400. doi: 10.1111/biom.13062. Epub 2019 Jun 3. PMID 31009064
- [Derived] Jarskog LF, Hamer RM, Catellier DJ, Stewart DD, Lavange L, Ray N, Golden LH, Lieberman JA, Stroup TS; METS Investigators. Metformin for weight loss and metabolic control in overweight outpatients with schizophrenia and schizoaffective disorder. Am J Psychiatry. 2013 Sep;170(9):1032-40. doi: 10.1176/appi.ajp.2013.12010127. PMID 23846733
- [Derived] Khan AY, Macaluso M, McHale RJ, Dahmen MM, Girrens K, Ali F. The adjunctive use of metformin to treat or prevent atypical antipsychotic-induced weight gain: a review. J Psychiatr Pract. 2010 Sep;16(5):289-96. doi: 10.1097/01.pra.0000388624.91039.a3. PMID 20859106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blind, placebo-controlled multicenter trial conducted between March 2009 and February 2010 at 17 academic, veterans affairs, and private research clinics. 146 clinically stable overweight outpatients with chronic schizophrenia and schizoaffective disorder were enrolled.
Pre-assignment Details: Prior to randomization prospective participants were screened for eligibility
Groups:
- Placebo: Matching over-encapsulated placebo pills
- Metformin: Metformin 500 mg pills over-encapsulated up to 4 pills daily as tolerated
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 71 | 75
Completed | 58 | 58
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 71 | 75 | 146
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (10.3) | 41.4 (11.5) | 43.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 49 | 52 | 101

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Body Weight Change Between Participants Assigned to Metformin and Participants Assigned to Placebo
Description: Mean difference in body weight change between participants assigned to metformin and participants assigned to placebo from baseline to last study visit (up to 16 weeks)
Time Frame: Measured at the last study visit
Population: Evaluable population that took assigned study treatment
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
kilograms | -1.0 [-2.0 to -0.0] | -3.0 [-4.0 to -2.0]

2. Secondary Outcome: Change in Total Cholesterol From Baseline to 16 Weeks
Description: Total cholesterol
Time Frame: 16 weeks
Population: randomized participants who took assigned treatment
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
mg/dL | 0.2 [-6.5 to 6.9] | -8.9 [-15.6 to -2.3]

3. Secondary Outcome: Change in HDL Cholesterol From Baseline to 16 Weeks
Description: high-density lipoprotein
Time Frame: 16 weeks
Population: randomized participants who took assigned treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
mg/dL | -0.4 [-2.3 to 1.4] | -0.6 [-2.4 to 1.2]

4. Secondary Outcome: Change in LDL Cholesterol From Baseline to 16 Weeks
Description: low-density lipoprotein
Time Frame: 16 weeks
Population: participants who took assigned treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
mg/dL | -2.0 [-7.7 to 3.7] | -7.1 [-12.6 to -1.5]

5. Secondary Outcome: Change in Triglycerides From Baseline to 16 Weeks
Description: serum triglycerides
Time Frame: 16 weeks
Population: participants who took assigned treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
mg/dL | 13.2 [-0.3 to 26.7] | -7.0 [-20.4 to 6.3]

6. Secondary Outcome: Change in Fasting Glucose From Baseline to 16 Weeks
Description: fasting blood glucose
Time Frame: 16 weeks
Population: participants who took assigned treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
mg/dL | -1.6 [-4.3 to 1.2] | -2.3 [-5.0 to 0.5]

7. Secondary Outcome: Change in Fasting Insulin From Baseline to 16 Weeks
Description: Fasting insulin
Time Frame: 16 weeks
Population: participants who took assigned treatment
Measure: Mean (95% Confidence Interval); unit: mU/L
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
mU/L | 5.5 [-1.7 to 12.6] | 1.6 [-5.5 to 8.6]

8. Secondary Outcome: Change in Hemoglobin A1c From Baseline to 16 Weeks
Description: glycosylated hemoglobin
Time Frame: 16 weeks
Population: participants who took assigned treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 71 | 75
percent | 0.01 [-0.04 to 0.06] | -0.06 [-0.11 to -0.01]

ADVERSE EVENTS:
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 7/71 | 3/75
Other Adverse Events (participants affected / at risk) | 33/71 | 40/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | Metformin (N=75)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Suicidality (Psychiatric disorders) | 1 (1) | 1 (1)
rule-out seizure (Nervous system disorders) | 0 (0) | 1 (1)
elective knee-surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exacerbation of schizophrenia (Psychiatric disorders) | 2 (2) | 0 (0)
rule-out myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | Metformin (N=75)
diarrhea (Gastrointestinal disorders) | 12 (12) | 25 (25)
headache (Nervous system disorders) | 17 (17) | 11 (11)
nausea (Gastrointestinal disorders) | 8 (8) | 12 (12)
Muscle pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (13)
abdominal discomfort (Gastrointestinal disorders) | 9 (9) | 12 (12)
weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
vomiting (Gastrointestinal disorders) | 3 (3) | 8 (8)

LIMITATIONS AND CAVEATS:
Changes over periods of more than 16 weeks are unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No